CLINICAL TRIAL: NCT06563089
Title: Hypoalbuminemia in Critically Sick Children at Assiut University Children's Hospital
Brief Title: Hypoalbuminemia in Critically Sick Children
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nada Mohamed Fathy, Resident Doctor, 71515, Assiut, Assiut University
Other Study IDs: Hypoalbuminemia
Record Dates: First submitted 2024-08-17; First posted 2024-08-20 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Hypoalbuminemia
MeSH Terms: conditions — Hypoalbuminemia | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: blood sampling — Albumin level in blood

SUMMARY:
The primary outcome in this Hospital-based study is to correlate the significance of hypoalbuminemia with different prognosis and outcome of different pediatric diseases.

The secondary outcomes of this study are i) to investigate the frequency of occurrence of hypoalbuminemia ii) to evaluate whether hypoalbuminemia on admission is a marker of adverse outcome in this population iii) whether correction of albumin by Human Albumin infusion or FFP helps in decreasing the length of stay in pediatric care unit, morbidity (e.g., duration of ventilator use) or mortality of the sick child.

DETAILED DESCRIPTION:
Serum albumin plays an essential role by maintaining intravascular oncotic pressure and facilitating the transport of many hormones, drugs and bioactive elements in blood circulation. Furthermore, several previous studies showed other functions of albumin such as antioxidant effects, inhibition of platelet aggregation, anti-inflammatory and anti-apoptotic effects. Hypoalbuminemia is a frequent and early biochemical derangement in critically ill-patients. Hypoalbuminemia was defined as an albumin level of less than 3.4 g/dL for patients 7 months or older and less than 2.5 g/dL for patients younger than 7 months. Awais et al. categorized hypoalbunemia to mild hypoalbuminemia (patients with serum albumin levels of 3.3 to 3.4 g/dL), mild-moderate hypoalbuminemia (serum albumin levels of 3.1 to 3.2 g/dL), moderate-severe hypoalbuminemia (serum albumin levels of 2.8 to 3.0 g/dL) and severe hypoalbuminemia (serum albumin levels of 1.2 to 2.7 g/dL). The etiology of hypoalbuminemia is complex. In general, it is ascribed to diminished synthesis in malnutrition, malabsorption and hepatic dysfunction or increased losses in nephropathy or protein-losing enteropathy. Inflammatory disorders can accelerate the catabolism of albumin, while simultaneously decreasing its production. Diversion of synthetic capacity to other proteins (acute-phase reactants) is another likely cause of hypoalbuminemia in critically ill-patients. During critical illness, capillary permeability increases dramatically and alters albumin exchange between intravascular and extravascular compartments. Hypoalbuminemia in patients is a marker of disease severity and has been associated with prolonged ventilatory dependence and length of intensive care stay. It is also an independent predictor of mortality and it is associated with poor outcome in critically ill-patients. There is a paucity of data evaluating serum albumin levels and outcome of critically ill-children admitted to intensive care unit (ICU). The goal will be to evaluate whether hypoalbuminemia on admission is a marker of adverse outcome.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with an albumin level of less than 3.4 g/dL for patients 7 months or older and less than 2.5 g/dL for patients younger than 7 months.
2. Patients with Severe sepsis, Respiratory diseases, Neurological diseases, Cardiac diseases, Blood diseases and gastrointestinal diseases with low albumin level .

Exclusion Criteria:

1. Immune deficiency patients
2. Malabsorption syndrome patients
3. Celiac disease patients
4. Protein loosing enteropathy patients
5. Nephrotic syndrome patients
6. Chronic liver disease patients

Ages: 1 Month to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: critically sick children with hypoalbuminemia
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2024-09-15 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
to correlate the significance of hypoalbuminemia with different prognosis and outcome of different pediatric diseases. 5 | Baseline
  To evaluate whether hypoalbuminemia is a predictor of adverse outcome in different disease

REFERENCES:
- [Background] Goldwasser P, Feldman J. Association of serum albumin and mortality risk. J Clin Epidemiol. 1997 Jun;50(6):693-703. doi: 10.1016/s0895-4356(97)00015-2. PMID 9250267
- [Background] Rady MY, Ryan T. Perioperative predictors of extubation failure and the effect on clinical outcome after cardiac surgery. Crit Care Med. 1999 Feb;27(2):340-7. doi: 10.1097/00003246-199902000-00041. PMID 10075059
- [Background] Fleck A, Raines G, Hawker F, Trotter J, Wallace PI, Ledingham IM, Calman KC. Increased vascular permeability: a major cause of hypoalbuminaemia in disease and injury. Lancet. 1985 Apr 6;1(8432):781-4. doi: 10.1016/s0140-6736(85)91447-3. PMID 2858667
- [Background] Horowitz IN, Tai K. Hypoalbuminemia in critically ill children. Arch Pediatr Adolesc Med. 2007 Nov;161(11):1048-52. doi: 10.1001/archpedi.161.11.1048. PMID 17984406
- [Background] Nicholson JP, Wolmarans MR, Park GR. The role of albumin in critical illness. Br J Anaesth. 2000 Oct;85(4):599-610. doi: 10.1093/bja/85.4.599. No abstract available. PMID 11064620
- [Background] Vincent JL, Dubois MJ, Navickis RJ, Wilkes MM. Hypoalbuminemia in acute illness: is there a rationale for intervention? A meta-analysis of cohort studies and controlled trials. Ann Surg. 2003 Mar;237(3):319-34. doi: 10.1097/01.SLA.0000055547.93484.87. PMID 12616115
- [Background] Zimmerman JE, Kramer AA, McNair DS, Malila FM. Acute Physiology and Chronic Health Evaluation (APACHE) IV: hospital mortality assessment for today's critically ill patients. Crit Care Med. 2006 May;34(5):1297-310. doi: 10.1097/01.CCM.0000215112.84523.F0. PMID 16540951
- [Background] Durward A, Mayer A, Skellett S, Taylor D, Hanna S, Tibby SM, Murdoch IA. Hypoalbuminaemia in critically ill children: incidence, prognosis, and influence on the anion gap. Arch Dis Child. 2003 May;88(5):419-22. doi: 10.1136/adc.88.5.419. PMID 12716714